CLINICAL TRIAL: NCT03723044
Title: Multistability: Perception is Inspired by Noise
Acronym: MUSPIN-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: GIPSA-LAB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.059
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: No Conditions
Keywords: Multistable Perception; Micro eye movement; Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Other: EEG and occulometry

INTERVENTIONS:
Other: EEG and occulometry — Each participants will spend two sessions of EEG and occulometry during a visual cognitive task where she/her will be presented with multi-stable visual stimuli to gaze at for one or two minutes. Depending on the experimental conditions, the participant will provide or not her/his perceptual state (i.e. which stimulus has been perceived ).

SUMMARY:
Some stimuli, such as sinusoidal networks in motion, or the best known, Necker's cube, are simple visual stimulations generating interpretations of unstable and oscillatory shapes or movements, mutually exclusive. Currently, the explanatory models of these perception phenomena are based on adaptation and learning mechanisms as well as the importance of noise in the perceptual and decision-making system. Often noise is a harmful component, but it can also be a facilitator in perceptual systems: the investigator's eye is always in motion, it is the micro-movements during eye fixation (phase of eye stability). In particular, the role of micro-eye movements has been identified in perceptual systems, and it will be necessary here to relate these micro-movements to the perceptive tilts facing multisable stimuli. However, how to access the perceptive states is a real question, since it has been shown that the participant's transfer of his perceptual state by means of a motor response can alter the very state of the percept. This is why the EEG activity will be analyzed to learn to discriminate the different percepts over time, without disruption of the participant's perceptual exploration endogenous activity.

DETAILED DESCRIPTION:
Each participant will benefit from a medical interview before inclusion to eliminate the contraindications to this study. The maximum duration of the individual participation of each subject in this study is 5 hours in two sessions. Each session lasts 2h30. Both sessions are spaced a maximum of 14 days apart. Each session includes EEG headset placement and oculometer calibration (20 min), followed by recording EEG and eye tracking activity during a visual cognitive task where the participant will be presented with multi-stable visual stimuli to watch. for one or two minutes after the tests. By repeating the essays and the conditions of presentation, each session will be organized in six blocks of 20 minutes each, interspersed with a break.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Medical examination carried out before the participation in the research
* Age between 18 and 55 years
* Minimum level of studies
* Obligation to join the social security system
* normal or corrected vision normal

Exclusion Criteria:

* Subject included in another clinical and / or therapeutic experimentation in progress
* Major vision disorder
* Past or current neurological or neuropsychiatric pathologies
* History of cranial trauma with loss of consciousness.
* Medication treatments likely to modulate brain activity: benzodiazepine, antidepressants, neuroleptics, lithium, etc.
* Diabetes, cardiac pathology, immunodeficiency.
* Medication treatments likely to modulate the activity of the cardiovascular system.
* History of abuse or recent ingestion of alcohol, hard drugs or doping products.
* Consumption of more than 15 cigarettes per day
* Subject deprived of liberty by a judicial or administrative decision (L1121-6 CSP)
* Major subject subject to a legal protection measure or unable to express their consent (L1121-8 CSP)
* Pregnant, parturient and nursing mothers (L1121-5)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Micro-eye movement | along the complete experiment (2 hours) per session and per participant.
  Eye movements will be recorded with an eye-tracker : the continuous gaze position at each sampling period (1ms)
Electroencephalography | along the complete experiment (2 hours) per session and per participant.
  EEG will be recorded with 64 scalp electrodes (sampling rate 1kHz) with alpha and gamma waveform to found synchronuous neural correlates with the peceptive changes.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No